CLINICAL TRIAL: NCT00464880
Title: A Randomized, Double-Blind, Parallel-Group, Cross-Over, 4-Period, 4 Treatment, Within-Subject Placebo-Controlled Study to Assess the Reno-Protective Effect of Renin Inhibition With Aliskiren as an Alternative to Irbesartan in Type 2 Patients With Incipient/Overt Diabetic Nephropathy
Brief Title: Effects of Aliskiren, Irbesartan, and the Combination in Hypertensive Patients With Type 2 Diabetes and Diabetic Nephropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2243
Record Dates: First submitted 2007-04-21; First posted 2007-04-24 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Diabetes Type 2
Keywords: Placebo-controlled study; assess the renoprotective effect of renin inhibition; Aliskiren as an alternative to irbesartan; Type 2 diabetes patients; incipient/overt diabetic nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aliskiren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aliskiren

SUMMARY:
This study will assess the reno-protective effect of renin inhibition with aliskiren as an alternative to irbesartan in type 2 diabetes patients with incipient/overt diabetic nephropathy.

DETAILED DESCRIPTION:
Antiproteinuric Effects of Aliskiren (Renin Inhibitor), Irbesartan (Angiotensin Receptor Antagonist) and the Combination in Hypertensive Patients With Type 2 Diabetes and Incipient/Overt Diabetic Nephropathy

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects between the ages of 30-80 years with a diagnosis of type 2 diabetes (World Health Organization criteria)
* Body mass index (BMI) within the range of 20 and 32.
* Incipient or overt diabetic nephropathy (urinary albumin excretion ≥ 100 but ≤ 2000 mg/day).
* Glomerular filtration rate (GFR) ≥ 40 ml/min documented in the last 4 months prior to randomization
* To be eligible for randomization, patients must fulfill the following criteria:

  1. Patients on ongoing hypertensive therapy must have a blood pressure ≥ 135/85 mmHg but lower than 170/105 mmHg at Visit 2 (Day -1) AND patients must be on stable antihypertensive medications for at least 8 weeks prior to Visit 2 (run-in period).
  2. Newly diagnosed hypertensive patients must have a blood pressure ≥ 135/85 mmHg but lower than 170/105 mmHg at Visit 2 (Day -1).
* Patients must be on stable hypoglycemic medications for at least 8 weeks prior to Visit 2 (Day -1).
* Patients must be willing and medically able to discontinue all angiotensin-converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB), aldosterone receptor antagonist and potassium sparing diuretic medications for the duration of the study.
* Female patients must be postmenopausal, have had a bilateral oophorectomy, or have been surgically sterilized or hysterectomized at least 6 months prior to screening.
* Oral body temperature within the range of 35.0-37.5 °C
* Able to provide written informed consent prior to study participation.
* Able to communicate well with the investigator and comply with the requirements of the study.

Exclusion Criteria:

* Severe hypertension, Grade 3 World Health Organization (WHO) classification (mean sitting diastolic blood pressure [MSDBP] ≥ 110 mmHg and/or mean sitting systolic blood pressure [MSSBP] ≤ 180 mmHg)
* Acetylsalicylic acid (ASA) treatment > 1 g/day or regular use of nonsteroidal anti-inflammatory drugs (NSAIDs)
* Kidney disease not caused by diabetes or hypertension
* Serum potassium < 3.5 or > 5.1 mEq/L
* GFR < 40 ml/min/1.73m2 as measured by the Modification of Diet in Renal Disease (MDRD) formula
* Serum albumin < 2.0 mg/dL
* History of hypertensive encephalopathy or cerebrovascular accident in the last 12 months prior to Visit 1
* Transient ischemic cerebral attack during the 6 months prior to Visit 1
* Current diagnosis of heart failure (New York Heart Association [NYHA] Class II-IV)
* History of myocardial infarction, unstable angina pectoris, coronary bypass surgery, or any percutaneous coronary intervention (PCI) during the 6 months prior to Visit 1
* Second or third degree heart block without a pacemaker
* Concurrent potentially life threatening arrhythmia or symptomatic arrhythmia
* Clinically significant valvular heart disease
* Type 1 diabetes mellitus
* Uncontrolled type II diabetes mellitus; hemoglobin subtype A1C (HbA1C) > 11%
* History of malignancy including leukemia and lymphoma (but not basal cell skin carcinoma) within the past five years
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulation.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
* Significant illness within the two weeks prior to dosing.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs including, but not limited to, any of the following:

  * History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection
  * Currently active or previously active inflammatory bowel disease during the 12 months prior to Visit 1
  * Currently active gastritis, duodenal or gastric ulcers, or gastrointestinal/rectal bleeding during the 3 months prior to Visit 1.
  * Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase
  * Evidence of hepatic disease, a history of hepatic encephalopathy, a history of esophageal varices, or a history of portacaval shunt
  * Current treatment with cholestyramine or colestipol resins
* History of immunocompromise, including a positive test result.
* History of a positive hepatitis B surface antigen (HBsAg) or hepatitis C test result.
* History of drug or alcohol abuse within the 12 months prior to dosing.
* Persons directly involved in the execution of this protocol.
* Any condition that, in the opinion of the investigator or the Novartis medical monitor, would jeopardize the evaluation of efficacy or safety
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol
* Known or suspected contraindications to the study medications, including history of allergy to ACE inhibitors and/or to thiazide diuretics or other sulfonamide derived drug
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study
* Use of any prescription drug or over-the-counter (OTC) medication which is prohibited by the protocol.
* Patients who previously participated in any aliskiren study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To investigate whether renin-inhibition using aliskiren 300 mg daily could be a treatment alternative to the angiotensin II receptor antagonist irbesartan 300 mg with an equivalent potential for reno-protection

SECONDARY OUTCOMES:
To investigate whether combination therapy using aliskiren 300 mg daily and irbesartan 300 mg daily has a greater effect on reno-protection than either drug alone
To investigate whether aliskiren, irbesartan or the combination reduce biomarkers of inflammation and cardiovascular risk

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Persson F, Rossing P, Reinhard H, Juhl T, Stehouwer CD, Schalkwijk C, Danser AH, Boomsma F, Frandsen E, Parving HH. Renal effects of aliskiren compared with and in combination with irbesartan in patients with type 2 diabetes, hypertension, and albuminuria. Diabetes Care. 2009 Oct;32(10):1873-9. doi: 10.2337/dc09-0168. Epub 2009 Jul 8. PMID 19587362